CLINICAL TRIAL: NCT04391543
Title: BIOpsychosocial Approach of the CAncer-RElated FAtigue
Brief Title: BIOpsychosocial Approach of the CAncer-RElated FAtigue (BIOCARE FActory)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Le Mans Universite (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MIP-2019-001; 2019-A02525-52 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2020-04-22; First posted 2020-05-18 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): 4 experimental session (baseline, after treatment, 6 month post treatment and 12 months post treatment) with :
  * comprehensive interview
  * cognitive tests
  * anthropometric measures
  * postural balance test
  * critical force test
  * Astrand-Ryhming test
  * self-questionnaire (QLQ-C30, FA12, Brief Cope et Hospital Anxiety and Depression Scale)
  * actimetry
  * clinical and biological characteristics
  * determination of inflammatory markers
  * skeletal muscle index
  Interventions: Other: Experimental session

INTERVENTIONS:
Other: Experimental session — * comprehensive interview
  * cognitive tests
  * anthropometric measures
  * postural balance test
  * critical force test
  * Astrand-Ryhming test
  * self-questionnaire (QLQ-C30, FA12, Brief Cope et Hospital Anxiety and Depression Scale)
  * actimetry
  * clinical and biological characteristics
  * determination of inflammatory markers
  * skeletal muscle index
  Other Names: Experimental Arm

SUMMARY:
One of the most common and stressful side effects of the disease and associated treatments is cancer-related fatigue. It deeply disrupts quality of life and can have a negative impact on patient survival. However, cancer-related fatigue is largely underestimated by patients and poorly taken into account by clinicians. One of the reasons for its poor management is a lack of knowledge of the underlying mechanisms and risk factors.

Although a multiplicity of factors are associated with the appearance of cancer-related fatigue, we do not know their respective share, nor the nature of their interactions. The phenomenon studied reveals complex and systemic interactions between the biological, psychological and social dimensions. Recent systematic reviews clearly identify 2 locks currently preventing a better understanding of the mechanisms of cancer-related fatigue: i) lack of longitudinal studies, ii) lack of interdisciplinary studies. It is precisely these two challenges that the BIOCARE FActory project wishes to respond to.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed at the Victor Hugo Clinic, Le Mans.
* Patients aged >or= 18 and < 80 years old at the time of inclusion
* Patients with a histologically proven primary breast cancer from stage I to IIIc
* Naive patient of anti-cancer treatment for this cancer
* Agreement to participate in the study by written, informed and signed consent of the patient
* Affiliated patients or beneficiaries of a social security scheme
* ECOG Performance Status score ≤ 2

Exclusion Criteria:

* Comorbidity which can explain the symptoms of fatigue (Long-term illness other than cancer, chronic fatigue syndrome)
* Breathing difficulties requiring the use of respiratory assistance
* Signs of polyneuropathy, amyotrophy or myasthenic syndrome
* Contraindications to physical exercise linked to heart failure.
* Treatment based on psychostimulants, psychotropics, antidepressants, antiepileptics or benzodiazepines for more than 3 months at the time of the study
* Presence or history of psychosis, bipolarity or severe depression
* History of stroke
* History of chronic fatigue
* History of musculoskeletal disorders of the lower limbs
* Pregnancy, breastfeeding
* Patient unable to undergo protocol monitoring for psychological, social, family or geographic reasons

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Sociability status | 18 months
  Change from baseline of a Comprehensive interview
Physical characteristics 1 | 18 months
  Change from baseline of height (in meters)
Physical characteristics 2 | 18 months
  Change from baseline of mass (in kilograms)
Physical characteristics 3 | 18 months
  Change from baseline of fat mass (in percentage)
Physical characteristics 4 | 18 months
  Change from baseline of leg volum
Postural stability | 18 months
  Change from baseline of maximum displacement speed of pressure centre at the postural stability test
Cognitive function 1 | 18 months
  Change from baseline of Stroop test score (higher score means worse outcome)
Cognitive function 2 | 18 months
  Change from baseline of Montreal Cognitive Assessment score (higher score means better outcome)
Cognitive function 3 | 18 months
  Change from baseline of Trail Making test score (higher score means worse outcome)
Fatigability | 18 months
  Change from baseline at critical force test measurement
Functional cardio-respiratory capability | 18 months
  Change from baseline of the maximum volum of oxygen during Astrand-Rhyming test
Quality of life status | 18 months
  Change from baseline of the European Organisation for Research and Treatment of Cancer quality of life C30 questionnaire score (higher score means better outcome)
Fatigue | 18 months
  Change from baseline of the European Organisation for Research and Treatment of Cancer Fatigue questionnaire score (higher score means worse outcome)
Anxiety | 18 months
  Change from baseline of the Hospital Anxiety and Depression scale score (higher score means worse outcome)
Emotional function | 18 months
  Change from baseline of the Brief Cope test score
Level of activity | 18 months
  Change from baseline of actimetry mesurement
Inflammatory status (pro-inflammatory cytokines) | 18 months
  Change from baseline of blood inflammatory markers determined by ELISA test (pro-inflammatory cytokines : IL-6, TNFα, IL-8, IL-1β)
Inflammatory status (anti inflammatory cytokine) | 18 months
  Change from baseline of blood inflammatory markers determined by ELISA test ( anti inflammatory cytokine : IL-1ra)
Sarcopenia 1 | 18 months
  Change from baseline of body masse index
Sarcopenia 2 | 18 months
  Change from baseline of musculo-skeletal index measurement on the third lumbar vertebra on scanner

CONTACTS AND LOCATIONS:
Overall Officials: Hugues Bourgeois, MD, Principal Investigator — Clinique Victor Hugo - LE MANS; Caroline Fonsegrive, MD, Principal Investigator — Centre Hospitalier du Mans
Locations (1):
- Le Mans University, Le Mans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leclercq A, Chatrenet A, Bourgeois H, Cojocarasu O, Mathie C, Martin T, Rahmani A, Morel B. Multidisciplinary analysis of cancer-related fatigue at the time of diagnosis: preliminary results of the BIOCARE FActory cohort. Support Care Cancer. 2024 Apr 30;32(5):319. doi: 10.1007/s00520-024-08520-4. PMID 38689167
- [Derived] Chartogne M, Rahmani A, Landry S, Morel B. Comparison of neuromuscular fatigability amplitude and etiologies between fatigued and non-fatigued cancer patients. Eur J Appl Physiol. 2024 Apr;124(4):1175-1184. doi: 10.1007/s00421-023-05347-5. Epub 2023 Nov 12. PMID 37952231
- [Derived] Chartogne M, Leclercq A, Beaune B, Boyas S, Forestier C, Martin T, Thomas-Ollivier V, Landry S, Bourgeois H, Cojocarasu O, Pialoux V, Zanna O, Messonnier LA, Rahmani A, Morel B. Building a biopsychosocial model of cancer-related fatigue: the BIOCARE FActory cohort study protocol. BMC Cancer. 2021 Oct 23;21(1):1140. doi: 10.1186/s12885-021-08831-3. PMID 34688272